CLINICAL TRIAL: NCT03016247
Title: Pilot Study Evaluating the Effects of a Trust-Building Intervention on Adolescent Weight Self-Management Behaviors
Brief Title: TRUST Study of Adolescent Weight Self-Management
Acronym: TRUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Heather K Hardin, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-16-49
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Adolescent Obesity
Keywords: magnetic resonance imaging, trust, reward
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): Group will receive a single visit with a Nutritionist for dietary and physical activity counseling
  Interventions: Behavioral: Enhanced Usual Care
- TRUST intervention (Experimental): Group will receive parent-adolescent trust-building and weight self-management training.
  Interventions: Behavioral: TRUST Intervention

INTERVENTIONS:
Behavioral: TRUST Intervention — The TRUST intervention will be guided by Rotenberg's Framework of Interpersonal Trust 3. The TRUST group will meet with an interventionist trained in weight self-management for eight 90-minute weekly sessions. Each session will include adolescent/parent trust-building exercises (honesty, reliability, emotional connection), didactic content, experiential skills developing (nutrition label reading), behavior-change goal-setting, and problem-solving.
  Other Names: Trust-building weight Self-management Together
  Arms: TRUST intervention
Behavioral: Enhanced Usual Care — Single meeting with a Nutritionist for physical activity and eating counseling.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of this pilot study is to evaluate the effect of the Trust-building weight Self-management Together (TRUST) intervention on weight self-management behaviors and neural processing in overweight/obese adolescents. Study aims include comparing the effects of the TRUST intervention with Enhanced Usual Care on BMI and quality of life in overweight/obese early adolescents and exploring differences in neural processing (DMT/TPN switching and reward activation).

DETAILED DESCRIPTION:
Background Adolescent obesity is a serious concern in the US, placing young people at risk for multiple chronic conditions. Family-based interventions are most effective with this challenge1, but adolescents' trust of their parents diminishes around age 14 as a result of developmental brain changes2-4. This distrust may thwart family-based weight self-management interventions; therefore, in this study the investigators will assess the effects of building trust between adolescents ages 10-12 and their parents, alongside weight self-management skills. Trust is a reciprocal quality between dyads that crosses the cognitive, affective, and behavioral domains and consists of honesty, receptivity to disclosures, and perceived compatibility between one's actions and words, which results in a sense of psychological safety from criticism, embarrassment, or harm.5 Because of its central role in adolescent-parent social interactions/relationships, trust may be a key factor in acquiring and sustaining healthy behaviors. Despite literature supporting the importance of interpersonal social interactions in making behavior change1,6, no studies to date have simultaneously examined both the biological and behavioral pathways through which trust in interpersonal interactions elicits behavior change. Thus, we employ a study design that includes basic research on the role of trust as a putative intervention target for behavior change in the context of an ongoing experimental clinical study testing the effects of a family trust-building behavioral intervention designed to reduce BMI in overweight/obese adolescents. We posit that adolescent-parent trust is a unique and potentially important interpersonal communication putative target to engage behavior change to improve healthy eating, physical activity, and sleep in overweight/obese adolescents, which will in turn reduce BMI.

Research in the area of cognitive processing has identified two broad cortical neural networks, the Task Positive Network (TPN), which is involved with using skills, knowledge and self-monitoring for problem solving and goal-directed action, and the Default Mode Network (DMN), which focuses on emotion-management, self-awareness and relationships. Neural network activity is consistently observable on fMRI. These broad networks tend to be antagonistic, such that when one network is activated, the other is inhibited; this inhibition/activation of the two modes may have important implications for self-management efforts, since an individual can only efficiently adopt one mode-processing either tasks or emotions--at a given time.7,8 The Analytic v. Emotional network theory suggests that flexible and balanced activity between modes is optimal9-11 and may be modified by learning/training, including practices such as meditation.12

In the work of one of the SMART Center Core leaders 7,13, Dr. Anthony Jack, fMRI revealed that individuals, when presented with an analytical (mechanical) problem, tended to activate analytic processing while deactivating empathic (emotional) processing. Conversely, when presented with a social problem, individuals tended to deactivate the analytic processing pathways in favor of increased emotional processing. These compelling findings provide an intriguing new way to examine an individual's approach to health behaviors and provide a new view into the brain-behavior connection. Jack's work 14,15 has shown that "coaching" exerts a dose-dependent effect on brain regions associated with motivation. In particular, focused training increased activity in the ventral-medial prefrontal cortex (VMPFC in left side of Figure 2) and adjacent regions of sub-genual anterior cingulate and nucleus accumbens. These regions, which are part of the default mode network, are implicated in motivation. In addition to identifying differences in brain function and connectivity,15 we are also examining any structural changes in brain anatomy brought about by the interventions. These are hypothesized to occur in the same regions as functional changes.16,17 Prior studies have demonstrated that residual activity in the DMN, during the performance of tasks sub served by the TPN, causes errors and lapses of attention.18,19 On the other hand, the DMN plays a key role in social cognition and motivation, specifically the generation of affective meaning 15,20,21 or purpose in life. A key hypothesis is that effective tuning of DMN function is essential for effective TPN function, which is required for successful self-management. Although neural and cognitive capacities which underlie self-management behavior may be non-specific in nature, identifying key mechanisms and signatures of effective interventions will better inform theoretical frameworks of self-management science.

Significance Our premise is that self-management interventions that target both analytic and emotional components of neurocognitive processing will be most effective in helping individuals achieve self-management outcomes. We are using functional magnetic resonance imaging (fMRI) to examine the relationship between two large-scale cortical networks, the default mode network (DMN) and the task positive network (TPN), and their contributions to behavior. Numerous studies have demonstrated that these networks may suppress each other, as measured both during task performance and in the resting state, which represents a marker of psychological health 22. The investigators interpret these findings as the ability to flexibly move between distinct cognitive modes associated with each network 13. A key hypothesis is that effective tuning of DMN function is essential for effective TPN function, and in turn, optimal performance of self-management activities. We posit that the TRUST intervention will influence the adolescent's emotional (DMT) neural processing through the trust-building component, while the analytic (TPN) neural processing will be influenced by the skills building component of the intervention, both of which work together to promote healthy weight self-management behaviors 23. In addition, the investigators hypothesize that the TRUST intervention will influence the adolescent's neurological reward activation between social reward and palatable food reward demonstrated in the ventral striatum 24,25.

As demonstrated in our model-consistent with the P30 Center of Excellence in Self-Management Research (SMART) framework being used for all SMART Center studies-the investigators hypothesize that an adolescent's weight self-management behaviors are influenced by the ability of the individual to balance DMT and TPN neural processing. the investigators posit that a reduction of body mass index (BMI) and an improvement in quality of life (QOL) will result from weight self-management behaviors (eating, physical activity, sleep) as mediated by two neural processes (DMT/TPN task-switching, reward activation), adolescent trust of parent, parent trust of adolescent, adolescent/parent relationship quality, social support, decision-making, self-efficacy, patient activation, and self-regulation. The influence of potential moderators (gender, binge-eating, perceived stress, depressive symptoms, executive functioning, parenting style) will be assessed for their effect on the relationship between the intervention and the proximal and distal outcomes. The investigators will conduct a two-group intervention trial to describe the effects of the TRUST intervention on BMI, QOL, and cognitive task switching between the DMT and TPN neural networks.

If the findings confirm the hypotheses, the intervention can serve as a model for improving adolescent weight self-management behaviors. The conduct of this project will also provide invaluable insights on the neurocognitive underpinnings of trust-building and its role as a facilitator of adolescent weight self-management. Specifically, the knowledge gained from this project will provide a foundational evidence on how trust-building in primary relationships can lead to enhanced states of self-management and reward sensitivity. Improvements in weight self-managements behaviors have shown to improve health outcomes. Successful weight self-management behaviors are associated with increased survival and decreased morbidity. If successful, this trust-building weight self-management will provide an acceptable and feasible self-management intervention that allows parents and adolescents to work together to improve the health and well-being of the family. In general, the potential benefits of this project outweighs the potential risks, and we have an experienced team of investigators and research staff that are prepared to address the minimal risks that may occur.

Purpose/Aims

The purpose of this pilot study is to evaluate the effect of the Trust-building weight Self-management Together (TRUST) intervention on weight self-management behaviors and neural processing in overweight/obese adolescents. The aims of this two-group randomized trial are to:

1. Compare the effects of the TRUST intervention with Enhanced Usual Care on BMI and QOL in overweight/obese early adolescents;
2. Determine the extent to which gender, binge-eating, perceived stress, depressive symptoms, executive functioning, and parenting style moderate the effect of TRUST on BMI and QOL;
3. Compare the effects of the TRUST intervention with Enhanced Usual Care on weight self-management behaviors (eating, physical activity, sleep);
4. Determine the extent to which gender, binge-eating, perceived stress, depressive symptoms, executive functioning, and parenting style moderate the effect of TRUST on weight self-management behaviors (eating, physical activity, sleep); and
5. Explore differences in neural processing (DMT/TPN task-switching, reward activation) in the TRUST intervention and Enhanced Usual Care group outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 10-12 year old Cleveland Metropolitan School District student
* identified as overweight or obese (BMI >85th percentile for age/sex during school screenings)
* able to read, speak, and understand the English language
* able to complete a self-administered questionnaire

Exclusion Criteria:

* taking medications that alter appetite or weight
* stage 2 hypertension or stage 1 hypertension with end organ damage
* severe behavioral problems that preclude group participation (as reported by parent/guardian)
* child involvement in another weight management program
* pregnancy
* family expectation to move from the region within 1 year

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 6 months
  Statistically significant change in BMI from baseline to 3 months and 6 months

SECONDARY OUTCOMES:
Eating | 6 months
  Change in Nutrient Data Systems Report data
Physical Activity | 6 months
  Change in accelerometer data
Sleep | 6 months
  Change in PROMIS-Sleep 4 scale score and Pediatric Daytime Sleepiness Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Heather K Hardin, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared for further analysis after main results are published.

REFERENCES:
- [Background] Heinberg LJ, Kutchman EM, Berger NA, Lawhun SA, Cuttler L, Seabrook RC, Horwitz SM. Parent involvement is associated with early success in obesity treatment. Clin Pediatr (Phila). 2010 May;49(5):457-65. doi: 10.1177/0009922809337531. Epub 2009 Jun 1. PMID 19487764
- [Background] Steinberg L. A Social Neuroscience Perspective on Adolescent Risk-Taking. Dev Rev. 2008 Mar;28(1):78-106. doi: 10.1016/j.dr.2007.08.002. PMID 18509515
- [Background] Jack AI, Dawson AJ, Begany KL, Leckie RL, Barry KP, Ciccia AH, Snyder AZ. fMRI reveals reciprocal inhibition between social and physical cognitive domains. Neuroimage. 2013 Feb 1;66:385-401. doi: 10.1016/j.neuroimage.2012.10.061. Epub 2012 Oct 27. PMID 23110882
- [Derived] Moore SM, Musil CM, Alder ML, Pignatiello G, Higgins P, Webel A, Wright KD. Building a Research Data Repository for Chronic Condition Self-Management Using Harmonized Data. Nurs Res. 2020 Jul/Aug;69(4):254-263. doi: 10.1097/NNR.0000000000000435. PMID 32205788